CLINICAL TRIAL: NCT04515953
Title: A Phase I Dose-escalation Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of a Single Administration of Extended-Release Injectable Suspension (ND-340) as Post-operative Analgesia in Patients With Total Knee Arthroplasty (TKA)
Brief Title: A Phase I Dose-escalation Study of a Single Administration of Extended-Release Injectable Suspension (ND-340)
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: pending
Sponsor: Nang Kuang Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QCR19001
Record Dates: First submitted 2020-07-08; First posted 2020-08-17 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-10

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Intervention Model Description: The first two arms of the placebo control and the 1st dose level ND-340 were randomly paralleled and then subsequently arms for ND-340 dose escalations.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Standard practice of pain management for post-TKA
  Interventions: Drug: IV-PCA
- ND-340 (Experimental): ND-340 90mg~320mg at dose escalations
  Interventions: Drug: ND-340

INTERVENTIONS:
Drug: ND-340 — ND-340: Subjects will receive a single administration of ND-340 at the specified dose in each arm after TKA.
  Arms: ND-340
Drug: IV-PCA — IV-PCA: Intravenous patient-controlled analgesia (IV-PCA), morphine, will be administered in subjects of control group after TKA for postoperative pain management as standard practice.
  Arms: Control

SUMMARY:
This study focused on ND-340 extended release injection suspension for patients undergoing total knee arthroplasty with a one-time nerve blockade to assess drug side effects, pharmacokinetics and the effect of pain relief after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with age between 20 and 80 (inclusive) years old at the screening visit
2. With physician's order to undergo scheduled primary unilateral TKA
3. Female subject with childbearing potential must have a negative serum pregnancy test at the screening visit
4. Both male and female subjects with childbearing potential must agree to use 2 medically accepted methods of contraception (e.g., barrier contraceptives [male condom, female condom, or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], and intrauterine devices) during the course of the study with their partners (excluding women who are not of childbearing potential and men who have been sterilized).
5. Able and willing to comply with all study visits and procedures
6. Able to speak, read, and understand the language of the informed consent form (ICF), study questionnaires, and other instruments used for collecting subject-reported outcomes, in order to enable accurate and appropriate responses to pain scales and other required study assessments
7. Willing and capable of providing written informed consent

Exclusion Criteria:

1. Body weight < 50 kilograms or a morbidly obese (body mass index ≥ 35kg/m2)
2. Subject with American Society of Anesthesiologists (ASA) physical status > 3 at the screening visit
3. Undergoing or is plan to undergo bilateral or revision total knee replacement
4. Previous contralateral TKA or open knee surgery on the knee being considered for TKA in this study within 1 year prior to screening. Prior arthroscopy at least 1 week prior to TKA is permitted.
5. Use of any of the following medications within the time specified before TKA

   * Use of any opioid within 24 hours or long-acting opioid within 3 days
   * Use of any NSAID including selective COX-2 inhibitor within 3 days
   * Use of any selective serotonin reuptake inhibitors (SSRIs), gabapentin, pregabalin (LYRICA®), or duloxetine (CYMBALTA®) within 3 days
   * Use of monoamine oxidase inhibitors (MAOIs) within 14 days
6. Concurrent painful physical condition, diseases or concurrent surgery that may require analgesic treatment (such as NSAIDs or opioids) in the post-operative period for pain that is not strictly related to the surgery, and which may confound the post-operative assessments (e.g., significant pain from other joints including the non-index knee joint, chronic neuropathic pain, concurrent or prior contralateral TKA, concurrent foot surgery)
7. Pre-operative liver insufficiency as defined by liver function tests [i.e. alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), or total bilirubin] ≥ 1.5 times the upper limit of normal (ULN) at the screening visit
8. Pre-operative renal insufficiency (creatinine clearance < 60 mL/min) at the screening visit
9. Known of active infection with HIV, HBV, or HCV at the screening visit
10. With abnormal ECG at screening and admission, which is not suitable to participate into this study as judged by the investigator before TKA
11. With abnormal results of sensory examination as judged by the investigator before TKA
12. Administration of an investigational drug within 30 days or 5 elimination half- lives of such investigational drug, whichever is longer, prior to study drug administration; or planned administration of another investigational product or procedure during the study period
13. Receiving other surgeries within 30 days prior to screening
14. Receiving blood transfusion within 30 days prior to screening
15. With a history of allergy or hypersensitivity to local anesthetics
16. Previous hypersensitivity to or contraindication to any of the pain-control agents planned for surgical or post-operative use in this study (i.e., morphine, bupivacaine, tramadol, and acetaminophen)
17. History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years prior to screening
18. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that could interfere with study assessments or compliance in the opinion of the investigator
19. Current or historical evidence of any clinically significant disease or condition, especially terminal stage cancer, poorly controlled diabetic mellitus (i.e., HbA1c > 8%), or neurological disease that, in the opinion of the investigator, may increase the risk of study treatment and TKA, or complicate the subject's post-operative course or interfere with the determination of pain intensity related solely to the TKA
20. Subject with severe heart diseases (NYHA class-III and IV), with ischemic heart diseases (angina pectoris and myocardial infarction) and subject who underwent percutaneous transluminal coronary angioplasty (PTCA) or had treatments for coronary artery bypass graft within 6 months prior to screening
21. With pre-existed psychiatric or neurological deficits, which may compromise the neurological toxicity evaluations in this study by the investigator's judgment
22. With stroke within 1 year prior to screening
23. With bone cancer within 5 years prior to screening
24. Inability to understand or operate the PCA machine
25. Female subject who is breast-feeding, pregnant, or planning to become pregnant

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | up to 3 months
  The AEs of special interest, including any symptom of local anesthetic systemic toxicity (LAST), cardiac events, neurologic events, and falls, will be analyzed by cohort.
Cmax | 0(Pre-dose), 0.25, 0.5, 1, 1.5, 2, 4, 8, 18, 24, 32, 44, 56, 68, 80, 92,104,116,128,140,164 hour
  Maximum Plasma Concentration of ND-340
Tmax | 0(Pre-dose), 0.25, 0.5, 1, 1.5, 2, 4, 8, 18, 24, 32, 44, 56, 68, 80, 92,104,116,128,140,164 hour
  Time of peak concentration of ND-340
AUC 0-t | 0(Pre-dose), 0.25, 0.5, 1, 1.5, 2, 4, 8, 18, 24, 32, 44, 56, 68, 80, 92,104,116,128,140,164 hour
  Area under the plasma concentration versus time curve from zero to t of ND-340
AUC 0-∞ | 0(Pre-dose), 0.25, 0.5, 1, 1.5, 2, 4, 8, 18, 24, 32, 44, 56, 68, 80, 92,104,116,128,140,164 hour
  Area under the plasma concentration versus time curve from zero to infinity of ND-340
T1/2 | 0(Pre-dose), 0.25, 0.5, 1, 1.5, 2, 4, 8, 18, 24, 32, 44, 56, 68, 80, 92,104,116,128,140,164 hour
  Terminal half life of ND-340
CL/F | 0(Pre-dose), 0.25, 0.5, 1, 1.5, 2, 4, 8, 18, 24, 32, 44, 56, 68, 80, 92,104,116,128,140,164 hour
  Clearance/Bioavailability of ND-340
λz | 0(Pre-dose), 0.25, 0.5, 1, 1.5, 2, 4, 8, 18, 24, 32, 44, 56, 68, 80, 92,104,116,128,140,164 hour
  Terminal elimination rate constant
Vz/F | 0(Pre-dose), 0.25, 0.5, 1, 1.5, 2, 4, 8, 18, 24, 32, 44, 56, 68, 80, 92,104,116,128,140,164 hour
  Apparent volume of distribution during terminal phase after non-intravenous administration
MRT 0-∞ | 0(Pre-dose), 0.25, 0.5, 1, 1.5, 2, 4, 8, 18, 24, 32, 44, 56, 68, 80, 92,104,116,128,140,164 hour
  Mean residence time

SECONDARY OUTCOMES:
Pain intensity | up to 1 week
  The pain assessment in subjects will be analyzed by each cohort. The AUC of NRS-R or NRS-A within 24 hours (AUCNRS-R, 0-24 or AUCNRS-A, 0-24), 56 hours (AUCNRS-R, 0-56 or AUCNRS-A, 0-56), 80 hours (AUCNRS-R, 0-80 or AUCNRS-A, 0-80), 104 hours (AUCNRS-R, 0-104 or AUCNRS-A, 0-104), 128 hours (AUCNRS-R, 0-128 or AUCNRS-A, 0-128), and 164 hours (AUCNRS-R, 0-164 or AUCNRS-A, 0-164) after TKA will be analyzed and score-time curves will be plotted graphically.
The requirement for rescue pain medication | up to 1 week
  The requirement for rescuing pain medication will be analyzed by each cohort. Descriptive statistics will be used to analyze the percentage of subjects who use all IV-PCA morphine dose within 48 hours post-TKA or the percentage of subjects who use ULTRACET® within 7 days post-TKA, time period from the end of TKA to the first bolus dose of IV-PCA morphine or to the first use of ULTRACET® by cohort, the total amount of IV-PCA morphine administered within 48 hours post-TKA or the total amount of ULTRACET® administered within 7 days post-TKA.
The ambulation distance | up to 3 months
  The ambulation distance as measured by six-minute walk test (6MWT) at baseline and subsequent visits, and the change from baseline will be summarized descriptively by cohorts.
Range of motion of knee | up to 3 months
  The range of motion (ROM) of knee as measured by knee flexion and extension at baseline and subsequent visits, and the change from baseline will be summarized descriptively by cohorts.
WOMAC | up to 3 months
  The quality of life (QoL) as measured by WOMAC Index at baseline and subsequent visits, and the change from baseline will be summarized descriptively by cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Peng Lin, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Nang Kuang Pharmaceutical Co., LTD, Tainan, Taiwan (台灣), Taiwan